CLINICAL TRIAL: NCT06587945
Title: A Randomised Double-Masked Placebo-Controlled Trial of Nicotinamide Riboside Oral Supplementation in Macula Off Retinal Detachment
Brief Title: Nicotinamide Riboside Oral Supplementation in Macula Off Retinal Detachment
Acronym: NOMAD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Center for Eye Research Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NOMAD; U1111-1307-8530 (Other: Universal Trial Number, World Health Organisation)
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-07

CONDITIONS: Retinal Detachment
Keywords: Nicotinamide Riboside; Retinal detachment; Photoreceptors; Macula-off; Vitrectomy
MeSH Terms: conditions — Retinal Detachment | interventions — nicotinamide-beta-riboside; Vitrectomy

STUDY DESIGN:
Intervention Model Description: Multi-centre participant- and assessor-masked placebo-controlled randomised superiority trial with two parallel groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nicotinamide Riboside (Experimental): Oral Nicotinamide Riboside intake from date of presentation: 2g daily for 4 weeks followed by 1g daily for 16 weeks postoperatively
  Interventions: Dietary Supplement: Nicotinamide Riboside; Procedure: Vitrectomy and Gas tamponade
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo; Procedure: Vitrectomy and Gas tamponade

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Oral Nicotinamide Riboside, 2g daily for 4 weeks followed by 1g daily for 16 weeks
  Arms: Nicotinamide Riboside
Other: Placebo — Matched placebo
  Arms: Placebo
Procedure: Vitrectomy and Gas tamponade — Standard of care Vitrectomy surgery for retinal reattachment

SUMMARY:
Retinal detachment occurs when fluid separates the retina (a thin, light sensing tissue) from its usual attachment at the back of the eye. If detached, these retinal cells lose their normal blood supply and begin to die, which is the primary cause of vision loss in retinal detachment. The 'macula' refers to the very centre of the retina, with the highest density of retinal cells, most responsible for vision. Significant vision loss occurs when this part of the retina becomes separated (termed a 'macula-off retinal detachment'). Typically, surgery is required to repair the retinal detachment.

Supporting the health of retinal cells at the macula may prolong their survival after detachment and their recovery postoperatively. Recent evidence has shown that boosting our nicotinamide adenine dinucleotide (NAD+) levels may improve the health of these cells and prolong their survival if detached. Oral Nicotinamide Riboside (NR) is converted into NAD+, and while not studied for macula-off retinal detachments, has been safely used in a range of other conditions. This study is designed to help evaluate the safety and tolerability of NR to help preserve vision in people diagnosed with macula-off retinal detachment.

This study drug is given as an oral supplement (tablet) at the time of retinal detachment diagnosis, and daily for 20 weeks thereafter. The drug aims to prolong survival of cells in the retina (and macula) and their recovery after surgery.

The long-term goal of this treatment is to reduce loss of vision after retinal detachment. The researchers will compare NR to a placebo (a look-alike substance that contains no drug) to see if NR has a positive effect on photoreceptor survival and quality of vision postoperatively.

NR has been approved by the Therapeutic Goods Administration in Australia for many purposes but has not been approved for use in retinal detachment treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Able to give informed consent and comply with all study visits and procedures.
* Present within 10 days of macula-off retinal detachment (based on patient-reported history of loss of central vision)
* Present to the hospital with a visual acuity of hand motion or better in the study eye
* Have had previous cataract surgery in the study eye
* Have clinical indication for standard retinal reattachment surgery by means of a pars plana vitrectomy and gas tamponade
* In the opinion of the investigator, be able to safely undergo all study procedures.

Key exclusion Criteria:

* Any known significant ocular disease in the study eye (e.g., cornea opacity) which, in the opinion of the investigator, would preclude a visual acuity of at least 6/7.5 (20/25) following successful vitrectomy or limit adequate visibility of the retina.
* Any other ocular pathology in the study eye requiring treatment with topical ophthalmic drops or intravitreal injection.
* History of previous ocular surgery in the study eye other than uncomplicated cataract surgery with posterior chamber intraocular lens and intact posterior capsule or a refractive surgery (surgery must have occurred at least 3 months prior to the baseline visit).
* Participation in other clinical trials or use of any other investigational drugs or devices within 3 months prior to study participation.
* Females who are pregnant or lactating and women of childbearing potential.
* Known retinopathy, known hepatic disease (or history of significant chronic liver disease), or known renal disease. Patients Participants with diabetes and no known retinopathy may be enrolled.
* History of uncontrolled hypertension.
* History of stroke, transient ischemic attack, or major cardiac surgery within 3 months prior to study, or current treatment for systemic infection.
* Any ocular or systemic condition that in the opinion of the investigator could compromise the safety of the patientparticipant, or may interfere with the safety and tolerability assessments or study procedures of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Best-corrected Visual Acuity | 20 weeks postoperatively
Microperimetry | 20 weeks postoperatively
Contrast sensitivity | 20 weeks postoperatively

SECONDARY OUTCOMES:
Integrity of the photoreceptor layer on optical coherence tomography | 20 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: David Sousa, MD PhD FRANZCO, Principal Investigator — Center for Eye Research Australia
Locations (5):
- Australia (5):
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Cerulea, East Melbourne, Victoria
  - The Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
  - Dr David Fabinyi, Geelong, Victoria
  - Dr David Sousa, Geelong, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martens CR, Denman BA, Mazzo MR, Armstrong ML, Reisdorph N, McQueen MB, Chonchol M, Seals DR. Chronic nicotinamide riboside supplementation is well-tolerated and elevates NAD+ in healthy middle-aged and older adults. Nat Commun. 2018 Mar 29;9(1):1286. doi: 10.1038/s41467-018-03421-7. PMID 29599478
- [Background] Chen AC, Martin AJ, Choy B, Fernandez-Penas P, Dalziell RA, McKenzie CA, Scolyer RA, Dhillon HM, Vardy JL, Kricker A, St George G, Chinniah N, Halliday GM, Damian DL. A Phase 3 Randomized Trial of Nicotinamide for Skin-Cancer Chemoprevention. N Engl J Med. 2015 Oct 22;373(17):1618-26. doi: 10.1056/NEJMoa1506197. PMID 26488693
- [Background] Trammell SA, Schmidt MS, Weidemann BJ, Redpath P, Jaksch F, Dellinger RW, Li Z, Abel ED, Migaud ME, Brenner C. Nicotinamide riboside is uniquely and orally bioavailable in mice and humans. Nat Commun. 2016 Oct 10;7:12948. doi: 10.1038/ncomms12948. PMID 27721479
- [Background] Bai S, Sheline CT. NAD(+) maintenance attenuates light induced photoreceptor degeneration. Exp Eye Res. 2013 Mar;108:76-83. doi: 10.1016/j.exer.2012.12.007. Epub 2012 Dec 26. PMID 23274583
- [Background] Zhang X, Henneman NF, Girardot PE, Sellers JT, Chrenek MA, Li Y, Wang J, Brenner C, Nickerson JM, Boatright JH. Systemic Treatment With Nicotinamide Riboside Is Protective in a Mouse Model of Light-Induced Retinal Degeneration. Invest Ophthalmol Vis Sci. 2020 Aug 3;61(10):47. doi: 10.1167/iovs.61.10.47. PMID 32852543